CLINICAL TRIAL: NCT02245022
Title: Safety and Pharmacokinetics of Dolutegravir in Pregnant HIV Mothers and Their Neonates: A Pilot Study
Acronym: DolPHIN1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: ViiV Healthcare (Industry); Makerere University (Other)
Responsible Party: Principal Investigator, Catriona Waitt, Site sub-investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK12
Record Dates: First submitted 2014-09-12; First posted 2014-09-19 (Estimated); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: HIV; Pregnancy
Keywords: HIV; Prevention of mother to child transmission; Africa; Uganda; Pharmacokinetics; Pregnancy; Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — dolutegravir; Standard of Care; efavirenz; Lamivudine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dolutegravir 50mg od (Experimental): 30 patients who will receive dolutegravir 50mg once daily plus the same NRTI backbone as the active comparator group (lamivudine and tenofovir)
  Interventions: Drug: Dolutegravir 50mg od
- Standard of Care (Active Comparator): Patients randomised to receive antiretroviral therapy as per Uganda national guidelines (Efavirenz 600mg od based plus Tenofovir 300mg od and Lamivudine 300mg od)
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Dolutegravir 50mg od — Patients randomised to receive either Dolutegravir 50mg od or standard of care (Efavirenz 600mg od) plus Lamivudine 300mg od/ Tenofovir 300mg od
  Other Names: Tivicay (ViiV Healthcare); GSK1349572
  Arms: Dolutegravir 50mg od
Drug: Standard of Care — Patients are randomised 1:1 to receive either Dolutegravir 50mg once daily in combination with Lamivudine 300mg od and tenofovir 300mg od or standard of care (Efavirenz 600mg plus Lamivudine 300mg od and tenofovir 300mg od)
  Other Names: Efavirenz 600mg od; Lamivudine 300mg od; Tenofovir 300mg od
  Arms: Standard of Care

SUMMARY:
Aim: To evaluate dolutegravir (DTG) pharmacokinetics in pregnant HIV-infected women

Rationale: In developing countries many women present with a new HIV diagnosis in late pregnancy, and are at high risk of transmitting infection during delivery. Moreover, women may acquire NNRTI resistance from primary transmission, or use of nevirapine (NVP) in previous pregnancies. In these circumstances, DTG is likely to be more effective in reducing mother to child transmission of HIV than NNRTI-based regimens.

Study design: HIV positive pregnant women presenting with untreated HIV infection in late (≥28 -36 weeks gestation) pregnancy will be randomised 1:1 to receive DTG (50mg once daily) or standard of care (nevirapine or efavirenz) + 2 NRTIs. PK (0-24h) profile will be sampled in third trimester and post-partum.

Although this is primarily a PK study (and has been powered as such) randomisation is included to allow comparison of plasma HIV VL responses against standard of care (NVP or EFV) and is essential for evaluation of secondary endpoints of safety and efficacy of DTG in pregnancy.

Number recruited N=30 per group

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) in pregnancy is able to effectively reduce mother-to-child transmission (MTCT) of HIV. If untreated, the risk of transmission is around 25% (greater with high viral loads) but ART administered optimally during pregnancy may reduce this risk to 1-2%. In order to successfully prevent infection, ART should be started in the first or second trimester, and should reduce maternal plasma viral load to undetectable levels. Unfortunately throughout low-middle income countries, MTCT rates are unacceptably high with an estimated 430 000 newborn children infected annually. The main causes for this are undiagnosed or late diagnosis of maternal infection, suboptimal adherence to therapy and drug resistance, particularly in mothers who have previously received single dose nevirapine.

In sub-Saharan Africa (SSA), women frequently engage with health services late in pregnancy, and new HIV diagnoses in the third trimester (≥28 weeks of pregnancy) are not uncommon. Risk of MTCT is high, especially as NNRTI-based therapy takes a median of 2 months to significantly reduce the HIV viral load, making it unlikely that commencement of these drugs in late pregnancy will offer protection of the infant from intrapartum transmission.

Vertical transmission of HIV remains a significant challenge in developing countries and antiretroviral prophylaxis for PMTCT is an important tool towards elimination of paediatric infections. Between 2009 and 2010, coverage of antiretroviral prophylaxis for prevention of mother to child transmission was 42% and an estimated 1.48 million infants were born to women living with HIV (WHO 2010). Global efforts are geared towards improving access to antiretrovirals for PMTCT by simplifying antiretroviral treatment protocols while ensuring optimal outcomes for HIV-infected women and their children (WHO 2010; WHO 2012).

Under consolidated antiretroviral guidelines issued by the WHO in 2013, efavirenz-based ART is now recommended the preferred NNRTI option for HIV-1 infected patients, including among women of childbearing age and pregnant women (WHO 2013). In 2012, Uganda adopted the Option B+ strategy for PMTCT of HIV. Under this strategy, lifelong ART is offered to all pregnant ART naïve women irrespective of CD4 count with efavirenz-based ART as the preferred treatment option. However, the effectiveness of this regimen could be compromised in the event of large populations of women who may have been either exposed to single dose nevirapine in the past or among women with transmitted NNRTI resistance.

The justification for studying DTG in pregnancy includes:

1. Likely widespread availability of generic DTG in the coming years. The manufacturer has indicated its willingness to make DTG available in low income countries, and is currently engaging with generic manufacturers. Estimates from the Clinton Foundation suggest that generic manufacture of DTG will make this drug affordable either as an alternative first line, or else second line agent (Hill 2013). Clinical guidelines from the US and Europe currently rank INSTIs such as raltegravir and elvitegravir alongside NNRTIs as preferred first line agents. INSTIs may replace NNRTIs in first line regimens due to their good safety and toxicity profile, lower propensity for drug interactions, and superior efficacy. Large phase III RCTs comparing raltegravir (Rockstroh, Dejesus et al. 2013), elvitegravir (Sax, DeJesus et al. 2012) and dolutegravir (van Lunzen, Maggiolo et al. 2012) against efavirenz-based therapy have shown superior virological outcome at 48 weeks, faster time to undetectable viral load, lower incidence of adverse events, and fewer treatment discontinuations, and these findings have recently been confirmed in a meta-analysis (Messiaen, Wensing et al. 2013).
2. Low risk for serious drug-drug interactions. The potential for drug-drug interactions is significantly less for INSTIs compared with other antiretrovirals (relative risk compared with raltegravir: boosted protease inhibitors [RR = 4.96], non-nucleoside reverse transcriptase inhibitors [RR = 2.48](Patel, Abdelsayed et al. 2011). These are particularly important considerations for low/middle income country settings where adults with newly diagnosed HIV infection often present with tuberculosis, or during antenatal screening in late pregnancy. Here DTG may carry significant advantages over NNRTIs, and other INSTIs. In the absence of alternatives to rifampicin-based TB therapy, DTG and raltegravir exposures are only moderately reduced (Dooley, Sayre et al. 2013), compared to larger (50-90%) reductions in concentrations of boosted PIs, nevirapine and elvitegravir. Dolutegravir is metabolized by glucuronidation (UGT1A1) with some contribution from CYP3A.
3. Rapid viral load drop potentially beneficial in late diagnosis during pregnancy. In Sub-Saharan Africa, pregnant mothers tend to engage with health services later in pregnancy compared with Europe, and new HIV diagnoses resulting from universal testing at ≥28w gestation are frequent. DTG results in a very rapid reduction in viral load; median time to undetectable viral load in the SINGLE study was 28 days vs. 84 days with Atripla (P<0.0001) (Walmsley, Antela et al. 2012). Use of DTG may lower risk of mother-to-child transmission of HIV in late presenters. Although meta-analysis shows no increase in birth defects with maternal efavirenz (Ford, Mofenson et al. 2010), there has been recent suspicion of neurological toxicity in a large French registry (Sibiude, Madelbrot et al. 2013) and neurodevelopmental delay in a South African cohort (Westreich, Rubel et al. 2010)
4. Proven efficacy in patients with established drug resistance to other antiretrovirals. In most resource-poor settings, options for anti-retroviral therapy are limited (2011), and the emergence of HIV drug resistance gives cause for concern (Hedt, Wadonda-Kabondo et al. 2008; WHO 2012). In a cross-sectional study conducted among HIV-1 antiretroviral naïve patients in five African countries, the highest prevalence of transmitted resistance was observed in Kampala, Uganda 12.3% (22 of 179; 7.5-17.1) (Hamers, Wallis et al. 2011). In Malawi, the prevalence of primary drug resistance in new infections was 6.1% which is comparable with figures of ~3% for South Africa (Manasa, Katzenstein et al. 2012), and 5.7% for Zambia (Hamers, Siwale et al. 2010), with over half of all mutations conferring resistance to non-nucleoside reverse transcriptases (NNRTI) (Wadonda-Kabondo, Banda et al. 2012). Studies across Africa have shown that treatment response to NNRTIs in mothers and children exposed to nevirapine (particularly single dose) during pregnancy is blunted (Musiime, Ssali et al. 2009). In this context, a novel class of ARV which is safe, affordable and effective is an urgent need
5. Safety profile in pregnancy. DTG is classified as FDA pregnancy Category B. There are no adequate and well-controlled studies in pregnant women. Because animal reproduction studies are not always predictive of human response, and dolutegravir was shown to cross the placenta in animal studies, the manufacturer recommends that this drug should be used during pregnancy only if clearly needed (ViiV 2013).
6. Necessity of investigating DTG PK in pregnant women. Alongside the clinical and humanitarian imperative to provide effective treatment for preventing HIV transmission in pregnant mothers with NNRTI-resistant HIV, there is an equally important ethical imperative to establish the safety, efficacy and pharmacokinetics of DTG in pregnant mothers and their breastfed infants in SSA, especially given the implementation of WHO Option B+, and the potential for widespread use of DTG in the forseeable future. Previous experience suggests it is universally the case that pregnant women in SSA receive new antiretrovirals (ARV) ahead of any proper evaluation, and clinical studies (if undertaken at all) occur at a much later stage after many mothers and infants have been exposed.
7. Importance of undertaking the study in SSA. Any pivotal study if undertaken in developed countries would have limited generalizability to an African setting because i) ARVs tend to be initiated later in gestation in newly presenting pregnant women, ii) the standard of care across SSA is likely to be an efavirenz or nevirapine-based regimen iii) infant breastfeeding is recommended in the presence of ARVs ii) host factors such as BMI, ethnicity etc may impact on pharmacokinetics (PK) of ARVs.
8. Continued administration of DTG for 2 weeks post-partum (whilst breastfeeding) to characterize PK in non-pregnant state. Under standard of care, the infant will receive 6 weeks of nevirapine syrup, and would be exposed to the NNRTI/NRTI/NRTI combination received by the mother under standard of care. In this study, infants will be exposed DTG via the breastmilk for a 2 week period following birth. We believe this risk to be acceptable given the potential benefits. Furthermore, the risk is unlikely to exceed any potential risk of in utero exposure to DTG. Drug-drug interactions between directly administered NVP and DTG ingested via the breastmilk are unlikely to have clinical significance, although we will study this. The potential risks of breastfeeding are fewer than those of giving formula feeding during the two week period that mothers continue to receive DTG postpartum. Replacement of breast feeding with formula feeding during the first two weeks post-partum would be unethical due to the loss of the immune benefits of colostrum to the neonate, risks intrinsic to formula feeding in low resource settings and increased risk of HIV transmission if mixed feeding occurs (Teasdale et al, 2011) The potential risks of low-level ARV causing drug-resistance in the infant should the PMTCT fail exist for the standard of care NNRTIs and NRTIs; it is not anticipated that DTG will carry a greater risk but nevertheless this is best monitored within a clinical trial setting before widespread uptake without monitoring.

Study Design Open label randomized trial of DTG in late pregnancy. HIV+ pregnant women (untreated at ≥28w gestation will be randomized 1:1 to receive a DTG-based regimen compared with standard of care (regimen not containing INSTI).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Willing to participate,
* Women age 18 years and above
* Pregnant
* Untreated HIV infection in late pregnancy at ≥28 - 36 weeks gestation

Exclusion Criteria:

* Received antiretroviral drugs in previous 6 months
* Ever received integrase inhibitors
* Serum haemoglobin < 8.0 g/dl
* Elevations in serum levels of alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN) or ALT >3xULN and bilirubin >2xULN (with >35% direct bilirubin)
* eGFR < 50ml/min
* Active Hepatitis B infection, history or clinical suspicion of unstable liver disease, or subjects with severe liver disease (Class C by Childs-Hugh criteria)
* Severe pre-eclampsia (e.g. HELLP), or other pregnancy related events such as renal or liver abnormalities (e.g. grade 2 or above proteinuria, elevation in serum creatinine (above 2.5 x ULN), total bilirubin ALT or AST)
* Paternal non-consent (where disclosure to male partner has been made)
* Clinical depression or clinical judgement suggests increased risk of suicidality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saye H Khoo, PhD, MBChB, Principal Investigator — University of Liverpool; Mohammed Lamorde, PhD, MBChB, Principal Investigator — Infectious Diseases Institute, Makerere University
Locations (2):
- Desmond Tutu HIV Foundation, Cape Town, Western Cape, South Africa
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dickinson L, Walimbwa S, Singh Y, Kaboggoza J, Kintu K, Sihlangu M, Coombs JA, Malaba TR, Byamugisha J, Pertinez H, Amara A, Gini J, Else L, Heiberg C, Hodel EM, Reynolds H, Myer L, Waitt C, Khoo S, Lamorde M, Orrell C; DolPHIN-1 Study Group. Infant Exposure to Dolutegravir Through Placental and Breast Milk Transfer: A Population Pharmacokinetic Analysis of DolPHIN-1. Clin Infect Dis. 2021 Sep 7;73(5):e1200-e1207. doi: 10.1093/cid/ciaa1861. PMID 33346335
- [Derived] Waitt C, Orrell C, Walimbwa S, Singh Y, Kintu K, Simmons B, Kaboggoza J, Sihlangu M, Coombs JA, Malaba T, Byamugisha J, Amara A, Gini J, Else L, Heiburg C, Hodel EM, Reynolds H, Mehta U, Byakika-Kibwika P, Hill A, Myer L, Lamorde M, Khoo S. Safety and pharmacokinetics of dolutegravir in pregnant mothers with HIV infection and their neonates: A randomised trial (DolPHIN-1 study). PLoS Med. 2019 Sep 20;16(9):e1002895. doi: 10.1371/journal.pmed.1002895. eCollection 2019 Sep. PMID 31539371

RESULTS

PARTICIPANT FLOW:
Groups:
- Dolutegravir 50mg od: Patients who will receive dolutegravir 50mg once daily plus the same NRTI backbone as the active comparator group (lamivudine and tenofovir)
  Dolutegravir 50mg once daily: Patients randomised to receive either Dolutegravir 50mg once daily or standard of care (Efavirenz 600mg once daily) plus Lamivudine 300mg once daily/ Tenofovir 300mg once daily
- Standard of Care: Patients randomised to receive antiretroviral therapy as per Uganda national guidelines (Efavirenz 600mg once daily based plus Tenofovir 300mg once daily and Lamivudine 300mg once daily)
  Standard of Care: Patients are randomised 1:1 to receive either Dolutegravir 50mg once daily in combination with Lamivudine 300mg once daily and tenofovir 300mg once daily or standard of care (Efavirenz 600mg plus Lamivudine 300mg once daily and tenofovir 300mg once daily)
Period: Overall Study
Arm/Group | Dolutegravir 50mg od | Standard of Care
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dolutegravir 50mg od | Standard of Care | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 31 | 60
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 14 | 16 | 30
  South Africa | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: AUC0-24 of DTG in Pregnant Women in Third Trimester and 2 Weeks Postpartum
Description: Rich PK with sampling at t0, 1, 2, 4, 6, 8 and 24 hours relative to drug dose
Time Frame: In 3rd trimester and 2 weeks postpartum
Population: Not all participants on dolutegravir underwent the intensive pharmacokinetic sampling - hence the discrepancy in numbers.
  This related to the challenges of doing such a study in pregnancy and postpartum
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Groups:
- Postpartum: Same patients as in arm 1, but with the pharmacokinetic parameters measured postpartum.
Arm/Group | Dolutegravir 50mg od | Postpartum
Number analyzed (Participants) | 28 | 17
ng*h/mL | 35322 [19196 to 67922] | 40127 [22795 to 59633]

2. Primary Outcome: Cmax of Dolutegravir
Description: Maximum plasma concentration of dolutegravir in pregnancy vs postpartum
Time Frame: After 2 weeks of starting dolutegravir, and again 2 weeks after delivery
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- Dolutegravir 50mg Once Daily: 30 patients who will receive dolutegravir 50mg once daily plus the same NRTI backbone as the active comparator group (lamivudine and tenofovir)
  Dolutegravir 50mg od: Patients randomised to receive either Dolutegravir 50mg od or standard of care (Efavirenz 600mg od) plus Lamivudine 300mg od/ Tenofovir 300mg od
Arm/Group | Dolutegravir 50mg Once Daily | Postpartum
Number analyzed (Participants) | 28 | 17
ng/mL | 2534 [1462 to 3986] | 2899 [1397 to 4224]

3. Primary Outcome: Trough Concentration
Description: Concentration at 24 hours after dose, immediately prior to next dose) of dolutegravir
Time Frame: At 2 weeks after starting dolutegravir and again 2 weeks after delivery
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Groups:
- Dolutegravir 50mg Once Daily: 30 patients who will receive dolutegravir 50mg once daily plus the same NRTI backbone as the active comparator group (lamivudine and tenofovir)
  Dolutegravir 50mg once daily: Patients randomised to receive either Dolutegravir 50mg once daily or standard of care (Efavirenz 600mg once daily) plus Lamivudine 300mg once daily/ Tenofovir 300mg once daily
Arm/Group | Dolutegravir 50mg Once Daily | Postpartum
Number analyzed (Participants) | 28 | 17
ng/mL | 642 [188 to 3088] | 777 [348 to 1210]

4. Secondary Outcome: Number of Participants Reporting Severe Adverse Events During Study Period
Description: Safety questionnaires at every scheduled and unscheduled study visit Infant safety questionnaires at all post-partum visits Self-reporting
  Participants were reviewed for safety and tolerability after 7, 14 and 28 days on treatment, and after 56 days if delivery had not taken place. Following delivery, safety assessments were
Time Frame: From 7 days after start of treatment to 6 months postpartum
Population: Analysis of participants experiencing a pre-defined Severe Adverse Event
Measure: Number; unit: participants
Arm/Group | Dolutegravir 50mg od | Standard of Care
Number analyzed (Participants) | 29 | 31
participants | 2 | 1

5. Secondary Outcome: Percentage of Women in Each Arm With VL < 50 Copies/mL, and <400 Copies/mL at Delivery
Description: HIV viral load will be measured at enrollment into the study and at delivery
Time Frame: At delivery
Population: Number with HIV viral load < 50 copies/ mL at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50mg od | Standard of Care
Number analyzed (Participants) | 29 | 31
Participants | 21 | 12

6. Secondary Outcome: Cord:Maternal Plasma DTG Ratio
Description: A maternal blood sample and a cord blood sample will be taken at delivery to calculate the transplacental transfer of Dolutegravir
Time Frame: At delivery
Population: Participants in DTG arm who had cord and maternal blood sampling at delivery This is calculated by the ratio of drug in the cord blood to the maternal plasma - both samples were taken simultaneously
Measure: Median (Full Range); unit: Cord: Maternal blood ratio
Arm/Group | Dolutegravir 50mg od
Number analyzed (Participants) | 16
Cord: Maternal blood ratio | 1.21 [0.51 to 2.11]

7. Secondary Outcome: Maternal Plasma: Breastmilk DTG Ratio
Description: At the timepoints indicated, a single maternal blood sample and a sample of breast milk will be taken to measure Dolutegravir levels in both matrices and allow estimation of transmammary drug exposure
Time Frame: At 2 weeks postpartum, and 24 hours after final maternal dose
Population: Participants in DTG arm who underwent breastmilk pharmacokinetic sampling The ratio is calculated by comparing the concentration in breastmilk to that in maternal blood, so giving the milk: plasma ratio which is a standard measure of this outcome.
Measure: Median (Full Range); unit: Milk to plasma ratio
Arm/Group | Dolutegravir 50mg od
Number analyzed (Participants) | 17
Milk to plasma ratio | 0.03 [0.03 to 0.04]

8. Secondary Outcome: Infant DTG Levels
Description: Infants from the Dolutegravir arm (N=30) will be randomised 1:1:1 to return for PK sampling 1, 2 or 3 days after the mother has discontinued Dolutegravir and changed to Standard of Care treatment. All infants will have a single capillary blood sample (heel prick) taken at 2 weeks postpartum, and then at the time point they have been randomised to.
Time Frame: At maternal steady state (2 weeks postpartum) and at 1, 2 and 3 days after transfer to standard of care
Population: Infants of mothers in DTG arm who underwent pharmacokinetic sampling
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dolutegravir 50mg od
Number analyzed (Participants) | 17
ng/mL | 66.7 [21 to 654]

9. Secondary Outcome: Number and Severity of Adverse Events and Laboratory Abnormalities
Description: Laboratory test measured routinely up until 3 days after change to standard of care. In addition, patients will remain under follow-up until 6 months postpartum, and laboratory tests will be performed if clinically indicated at any point. The routinely measured 'safety bloods' in this study are Full Blood Count, Urea and Electrolytes including eGFR, Liver Function Tests including Alanine Aminotransferase and Bilirubin
Time Frame: Up to 3 days after change to standard of care, approximately 2 weeks after delivery
Population: Number of participants with abnormal biochemical or haematological parameters
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50mg od | Standard of Care
Number analyzed (Participants) | 29 | 31
Participants | 2 | 0

10. Secondary Outcome: Percentage of Subjects Who Discontinue Treatment Due to Adverse Events
Description: Mothers will be switched to standard of care at 2 weeks postpartum
Time Frame: Until 2 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50mg od | Standard of Care
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

11. Secondary Outcome: Percentage of Mother to Child Transmission of HIV
Description: Infant HIV testing by PCR will be undertaken at six weeks and six months of age, as per Uganda National Policy
Time Frame: 6 months postpartum
Population: Number with mother to child transmission of HIV
Measure: Count of Participants; unit: Participants
Arm/Group | Dolutegravir 50mg od | Standard of Care
Number analyzed (Participants) | 28 | 31
Participants | 0 | 0

12. Secondary Outcome: Pharmacogenomic Factors Influencing Transplacental and Breast Milk Transfer of Drug
Description: Frequency of relevant polymorphisms and association with drug concentrations
Time Frame: End of study
Population: This analysis was not undertaken for the following reason. DolPHIN-1 was designed as a pilot study to inform the design of a larger study with longer follow up. We obtained funding for DolPHIN-2 before DolPHIN-1 was complete, and in this we have included genome wide association survey of 250 mothers (125 per arm). Because this study has higher power to explore the pharmacogenomics, it was felt that undertaking this analysis in DolPHIN-1 would not add further useful information.
Groups:
- Dolutegravir 50mg od: 30 participants who will receive dolutegravir 50mg once daily plus the same NRTI backbone as the active comparator group (lamivudine and tenofovir)
- Standard of Care/ Efavirenz 600mg: 30 participants randomised to standard of care
Arm/Group | Dolutegravir 50mg od | Standard of Care/ Efavirenz 600mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Until 6 months postpartum
Description: Causality assessments were undertaken by a dedicated clinical pharmacist using the Liverpool Causality Assessment Tool.
  Grade >3 AEs summarised
Arm/Group | Dolutegravir 50mg od | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/31
Other Adverse Events (participants affected / at risk) | 2/29 | 2/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolutegravir 50mg od (N=29) | Standard of Care (N=31)
Low haemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Maternal malaria (Infections and infestations) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dolutegravir 50mg od (N=29) | Standard of Care (N=31)
Low haemoglobin (Blood and lymphatic system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT02245022/Prot_SAP_000.pdf